CLINICAL TRIAL: NCT03204162
Title: Optimizing Integration of CPR Feedback Technology With CPR Coaching for Cardiac Arrest
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: KidSIM Simulation Program (Network)
Collaborators: KidSIM-ASPIRE (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: REB15-2187
Record Dates: First submitted 2017-04-25; First posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Cardiopulmonary Resuscitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teams with no CPR Coach (No Intervention): This will be a standardized Resuscitation team with no CPR Coach
- Teams with CPR Coach (Experimental): This will be a standardized Resuscitation team where one member will be the CPR Coach and provide CPR Coaching to the team.
  Interventions: Other: CPR Coaching

INTERVENTIONS:
Other: CPR Coaching — Teams in the experimental arm will have a member of their team assigned to be the CPR Coach. This person will provide CPR Coaching in the form of feedback in CPR quality (depth, rate) to the CPR providers as well as provide guidance on time for defibrillation, etc.
  Arms: Teams with CPR Coach

SUMMARY:
There is significant data showing that the quality of CPR performed is quite poor. Recent studies have shown that when real-time visual corrective feedback is available to CPR providers, quality (compression depth and rate) improves.

Pilot work at John's Hopkins Children's Hospital indicates that providing a CPR Coach whose role it is to provide real-time coaching during cardiac arrest, further improves the quality of CPR. This study will assess the impact of a CPR Coach for improving CPR quality and CPR perception in a team of healthcare providers during simulated CPA.

DETAILED DESCRIPTION:
Cardiopulmonary resuscitation (CPR) is provided for thousands of children with cardiopulmonary arrests (CPA) each year in North America. The quality of CPR directly impacts hemodynamics, survival, and neurologic outcome following cardiac arrest. Well-trained healthcare providers consistently fail to perform CPR within established Heart and Stroke Foundation of Canada (HSFC) resuscitation guidelines. The poor quality of healthcare provider CPR adversely affects survival outcomes and quality of life in cardiac arrest survivors.

CPR feedback devices that provide real-time visual corrective feedback during CPA have become valuable tools to help to improve the overall quality of CPR. The cardiac arrest literature shows that although CPR feedback devices help to improve the overall quality of CPR, there is still substantial room for improvement. A recent multicenter study involving ten pediatric institutions led by the principal investigator of this project evaluated the impact of CPR feedback on CPR quality during simulated CPA5. This study demonstrated that the use of CPR feedback improved depth compliance by 15.4% and rate compliance by 40.1%. However, overall compliance with guidelines in the CPR feedback group was still under 40% for depth and under 75% for rate.

Data collected by this research team suggests that a variety of factors may influence the effectiveness of real-time CPR feedback. CPR providers interviewed after a simulated cardiac arrest report that they often are distracted by other events while providing CPR, are unable to clearly see the device, or have difficulty interpreting the visual display on the CPR feedback device. Additionally, many providers' perception of CPR quality is inaccurate, with providers consistently overestimating the quality of CPR provided during simulated CPA, even when using CPR feedback. This suggests a need to improve provider perception of CPR and provider awareness of the CPR feedback device.

To improve the quality of CPR the investigators propose the implementation of a standardized resuscitation team structure with a CPR coach. To date, there have been no studies describing the optimal team structure required for integration of CPR feedback defibrillators during CPA. In this study,the investigators propose the concept of a CPR coach, whose primary responsibility is to provide real-time coaching during cardiac arrest to improve the quality of CPR. Preliminary pilot work done in the intensive care unit at Johns Hopkins Children's Hospital suggests that use of a CPR coach improves the quality of CPR in comparison prior teams that functioned without a CPR coach. This study will assess the impact of a CPR Coach for improving CPR quality and CPR perception in a team of healthcare providers during simulated CPA.

ELIGIBILITY:
Inclusion Criteria:

* Team Members: (i) Pediatric healthcare providers: such as nurses, nurse practitioners, respiratory therapists and residents (pediatric, emergency medicine, anesthesia, family medicine); and (ii) Basic Life Support (BLS), Pediatric Advanced Life Support (PALS) or Advanced Cardiac Life Support (ACLS) certification within the past two years;
* Team Leaders: (i) Residents (Year 3 or 4) in pediatrics, family medicine, anesthesia, or emergency medicine training programs or fellows in pediatric emergency medicine, pediatric critical care or pediatric anesthesia subspecialty training programs; (ii) Attending physicians from pediatric intensive care, pediatric emergency medicine, general pediatrics; and (iii) PALS certification in the past two years or are PALS

Exclusion Criteria:

* Not BLS certified

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
CPR Depth | During simulation scenario -Day 1
  Proportion of 1 minute epochs of CPR with depth of 5cm to 6cm

SECONDARY OUTCOMES:
CPR Rate | During simulation scenario - Day 1
  Proportion of 1 minute epochs of CPR with rate of 100-120 beats per minute
Chest Compression Fraction | During simulation scenario - Day 1
  Percentage of time that compressions are provided during pulselessness
Perception of CPR Quality - Depth | Data collected immediately following the simulation session - Day 1
  Perceived quality of CPR depth will be collected by survey following the simulated cardiac arrest event. Survey data will be compared with measured quality of CPR depth from the defibrillator
Perception of CPR Quality - Rate | Data collected immediately following the simulation session - Day 1
  Perceived quality of CPR rate will be collected by survey following the simulated cardiac arrest event. Survey data will be compared with measured quality of CPR rate from the defibrillator
Perception of CPR Quality - Chest compression fraction | Data collected immediately following the simulation session -Day 1
  Perceived chest compression fraction will be collected by survey following the simulated cardiac arrest event. Survey data will be compared with measured chest compression fraction from the defibrillator
Adherence to Pediatric Advanced Life Support Guidelines | Day 1 (baseline performance)
  To assess clinical performance, the investigators will use a tool that assesses the team's performance during the simulated scenario. There will be no baseline performance measurement, and performance will be measured via retrospective video review after the simulation session is complete. Raters will be trained in the use of the Clinical Performance Tool (CPT). The tool scores items on a three point scale, with 0 = task not done, 1 = task done but not completely or 2 = task done correctly. The tool examines clinical performance specifically and not psychomotor performance. The CPT also accounts for tasks done in the incorrect sequence or done too late. This instrument has been found to produce valid data for clinical performance during PALS scenarios. For this current study, the version of this tool that will be used was modified slightly and validated in a previous multi centre trial carried out by this research team.
Airway Management Performance | Day 1 (Baseline performance)
  In order to assess airway management, the investigators will measure time to successfully intubate the manikin during the simulated scenario. There will be no baseline measurement, but rather just a report of the time to intubation during the one cardiac arrest simulation scenario (as collected by retrospective video review)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Cheng, MD, Principal Investigator — University of Calgary
Locations (5):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Columbia University Hospital, New York, New York
  - Hasbro Children's Hospital, Providence, Rhode Island
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng A, Brown LL, Duff JP, Davidson J, Overly F, Tofil NM, Peterson DT, White ML, Bhanji F, Bank I, Gottesman R, Adler M, Zhong J, Grant V, Grant DJ, Sudikoff SN, Marohn K, Charnovich A, Hunt EA, Kessler DO, Wong H, Robertson N, Lin Y, Doan Q, Duval-Arnould JM, Nadkarni VM; International Network for Simulation-Based Pediatric Innovation, Research, & Education (INSPIRE) CPR Investigators. Improving cardiopulmonary resuscitation with a CPR feedback device and refresher simulations (CPR CARES Study): a randomized clinical trial. JAMA Pediatr. 2015 Feb;169(2):137-44. doi: 10.1001/jamapediatrics.2014.2616. PMID 25531167
- [Background] Cheng A, Overly F, Kessler D, Nadkarni VM, Lin Y, Doan Q, Duff JP, Tofil NM, Bhanji F, Adler M, Charnovich A, Hunt EA, Brown LL; International Network for Simulation-based Pediatric Innovation, Research, Education (INSPIRE) CPR Investigators. Perception of CPR quality: Influence of CPR feedback, Just-in-Time CPR training and provider role. Resuscitation. 2015 Feb;87:44-50. doi: 10.1016/j.resuscitation.2014.11.015. Epub 2014 Nov 26. PMID 25433294